CLINICAL TRIAL: NCT06340646
Title: Washington University Participant Engagement and Cancer Genomic Sequencing Center (WU-PE-CGS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202106129; U2CCA252981 (NIH)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cholangiocarcinoma; Multiple Myeloma; Colon Cancer; Rectal Cancer
Keywords: Participant engagement; Genetic testing; Cholangiocarcinoma; Multiple Myeloma; Colorectal cancer; Underrepresented populations
MeSH Terms: conditions — Cholangiocarcinoma; Multiple Myeloma; Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Return of Genetic Results (No Intervention): Participants will undergo germline genomic sequencing as part of consenting to the WU-PE-CGS program.
  Participants will be given the option to receive the results from the genomic sequencing. After they consent to the study, the types of results available to them will be explained by research staff. Participants will be able to choose to receive: (1) no results, or any combination of (2) biomarker information from cancer cells, (3) inherited mutations related to cancer, and (4) inherited mutations related to other medical issues. These choices will be presented to them via a discussion with study staff with accompanying paper information
- Return of Genetic Results (Experimental): Participants will undergo germline genomic sequencing as part of consenting to the WU-PE-CGS program.
  Participants will be given the option to receive the results from the genomic sequencing. After they consent to the study, the types of results available to them will be explained by research staff. Participants will be able to choose to receive: (1) no results, or any combination of (2) biomarker information from cancer cells, (3) inherited mutations related to cancer, and (4) inherited mutations related to other medical issues. These choices will be presented to them via a discussion with study staff with accompanying paper information
  Interventions: Other: Return of Genetic Results: Biomarker information from cancer cells; Other: Return of Genetic Results: Inherited mutations related to cancer; Other: Return of Genetic Results: Inherited mutations related to other medical issues

INTERVENTIONS:
Other: Return of Genetic Results: Biomarker information from cancer cells — Participants will receive a novel return of results report that is tailored to their choices.
  Arms: Return of Genetic Results
Other: Return of Genetic Results: Inherited mutations related to cancer — Participants will receive a novel return of results report that is tailored to their choices.
  Arms: Return of Genetic Results
Other: Return of Genetic Results: Inherited mutations related to other medical issues — Participants will receive a novel return of results report that is tailored to their choices.
  Arms: Return of Genetic Results

SUMMARY:
The overall goal of the WU-PE-CGS is to build a rigorous, scientific evidence base for approaches that direct engagement of cancer patients and post-treatment cancer survivors as participants in cancer research, and to investigate the impact of directly engaging participants in decisions regarding returning of genomic results on participants' health and satisfaction. Participants in this study will be presented with the choice of types of genomic results to receive, and the Engagement Optimization Unit (EOU) will investigate the impact of this intervention on participant knowledge, expectations of benefit, personal utility, and decisional conflict.

ELIGIBILITY:
Eligibility Criteria:

* Patients with cholangiocarcinoma, multiple myeloma, or early onset colon or rectal cancer.

  * If diagnosed with multiple myeloma, must be African-American.
  * If diagnosed with colon or rectal cancer, must be African-American AND must be no older than 65 years old at the time of diagnosis.
  * At least 18 years old
  * Able to understand and willing to sign an IRB-approved written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Participant knowledge of clinical genetic testing | Through completion of follow-up (estimated to be 5 years)
  11-item, Likert scale. This scale has 5 points ranging from strongly agree to strongly disagree. 1=Strongly Agree, 2=Agree, 3=Neither Agree nor Disagree, 4=Disagree, 5=Strongly Disagree for items (4, 6-11) are scored such that 'strong disagree' reflects a correct response and 'somewhat disagree' reflects a less confident correct response in the correct direction. Negatively worded items (items 1, 2, 3, and 5) are reverse scored so that 'strongly agree' reflects a correct response and 'somewhat agree' reflect a less confident response in the correct direction. This will be scored by adding up the numbers for each of the 11 items regarding participant knowledge of clinical genetic testing. The total score ranges from 5 to 55. A higher score for the participant represents higher participant knowledge.
Participant expectations of benefit | Through completion of follow-up (estimated to be 5 years)
  Participants will rate their expectation for 6 potential benefits of cancer genomic sequencing on a 4-point scale ranging from extremely unlikely to extremely likely. . 1=Strongly Agree, 2=Agree, 3=Disagree, 4=Strongly Disagree. This will be scored by adding up the numbers for each of the 8 items regarding participant expectations of benefit. The total score ranges from 6 to 24. A higher score for the participant represents higher levels of expectations.
Participant personal utility | Through completion of follow-up (estimated to be 5 years)
  Participant personal utility will be measured on a 7-point scale ranging from not at all useful to extremely useful. 1=Not at all useful, 2=A little useful, 3=Somewhat useful, 4=Neutral, 5=Useful, 6=Very useful, 7=Extremely useful. This will be scored by adding up the numbers for each of the 14 items regarding participant personal utility. The total score ranges from 14 to 98. A higher score for the participant represents higher personal utility.

SECONDARY OUTCOMES:
Participant anxiety | Through completion of follow-up (estimated to be 5 years)
  Participant anxiety will be measured using a 5-point Likert scale ranging from not at all to very much. 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much. This will be scored by adding up the numbers for each of the 6 items regarding participant cancer worry. The total score ranges from 0 to 24. A higher score for the participant represents higher participant cancer worry.
Participant satisfaction | Through completion of follow-up (estimated to be 5 years)
  Satisfaction will be measured using a 5-point Likert scale ranging from extremely satisfied to not at all. 1=Not at all satisfied, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Extremely satisfied. The total score ranges from 1 to 5. A higher score for the participant represents higher participant satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Colditz, M.D., DrPH, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share all data, software and know-how generated during the course of this work, without limitations except as prevented by prior agreement. This will include both the final datasets, as well as the data necessary to complete the aims. Will disseminate results from this research through presentations at public lectures, scientific institutions and meetings, and/or publication in major journals. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. Wherever applicable, data will be deposited to appropriate public repositories.
  All participants whose genomic data are collected will be consented for broad data sharing, and their genomic data will be included in the study deposits. Data documentation and de-identified data will be deposited for sharing along with phenotypic data, which includes demographics and diagnosis, consistent with applicable laws and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: The investigators agree to deposit data into database of Genotypes and Phenotypes (dbGaP) repository after data cleaning and quality control as soon as possible but no later than within three months, or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier. When data are released from dbGaP, the data will be made available to the Genomic Data Commons (GDC).
Access Criteria: The investigators agree that they will identify where the data will be available (dbGaP and GDC) and how to access the data in any publications and presentations that they author or co-author about these data, as well as acknowledge the repository and funding source in any publications and presentations. As they will be using the database of Genotypes and Phenotypes (dbGaP), which is an NIH-funded repository, this repository has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu